CLINICAL TRIAL: NCT06412757
Title: Silexan in the Treatment Of Posttraumatic Stress Disorder (STOP) Trial
Brief Title: Silexan in the Treatment Of Posttraumatic Stress Disorder Trial
Acronym: STOP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Deakin University (Other)
Collaborators: University of Melbourne (Other); Ramsay Clinic Albert Road (Unknown)
Responsible Party: Principal Investigator, Gregory Roebuck, Principal Investigator, Deakin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29307; HT9425-23-1-0885 (Other Grant/Funding Number: US Department of Defense CDMRP Contract Number)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: posttraumatic stress disorder; adjunctive treatment; Silexan; phytoceutical; pharmacotherapy; randomized controlled trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: The trial is a phase 3, 12-week, parallel-arm, randomized, placebo-controlled, double-blind trial. Participants will be randomly allocated to receive either (a) Silexan 160 mg or (b) an identical appearing inert placebo, daily for 12 weeks in addition to their usual prescribed medications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members will be blinded to allocation. Blinding will be maintained by ensuring that the packaging, appearance and color of the Silexan (treatment) and placebo capsules are identical. Placebo capsules will also include a sub-therapeutic amount of lavender oil to match the odour of the Silexan capsules. In addition, blinding will be maintained by identifying participants using anonymous participant identifier numbers; an independent statistician will coordinate randomization and an independent pharmacist will store and provide blinded batches to study team members for dispensing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silexan 160 mg (Experimental): Participants in the Silexan arm will take Silexan 160 mg daily in the morning for 12 weeks in addition to their usual prescribed psychoactive medications. Participants will be followed up at 2, 4, 6, 8 and 12 weeks of the intervention period, as well as at 4 weeks post-treatment (off-treatment follow-up period).
  Interventions: Drug: Silexan
- Placebo (Placebo Comparator): Participants in this arm will take two placebo capsules daily in the morning for 12 weeks in addition to their usual medications. Participants will be followed up at 2, 4, 6, 8 and 12 weeks of the intervention period, as well as at 4 weeks post-treatment (off-treatment follow-up period).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Silexan — Participants in the Silexan arm will take two over-encapsulated capsules, each containing 80 mg Silexan, daily orally in the morning in addition to their usual medications. No modifications of allocated interventions will be made for any trial participants; if appropriate (i.e following the emergence of adverse events) participants will be withdrawn from the intervention.
  Arms: Silexan 160 mg
Other: Placebo — Participants in the placebo arm will take two capsules containing an inert placebo daily orally in the morning in addition to their usual medications. The placebo capsules will contain a sub-therapeutic amount of lavender oil to mimic the odor of the experimental drug (Silexan).
  Arms: Placebo

SUMMARY:
Posttraumatic stress disorder (PTSD) is a common and debilitating mental illness. Current treatments for PTSD include psychotherapy and antidepressant medications. Many patients are unable to tolerate psychotherapy for PTSD and drop out of it. In addition, its effectiveness is limited. Up to 50 percent of patients who receive psychotherapy do not benefit from it. Antidepressant medications have only small benefits in PTSD. They also have unpleasant side effects that can make patients unwilling to take them. There is an urgent need to develop new treatments for PTSD that work and are well-tolerated. Silexan has the potential to provide an important alternative treatment for PTSD.

Silexan is derived from lavender oil. It is taken orally in the form of capsules. It is currently available over-the-counter in 14 countries, including Australia and the United States. Previous research has shown that it is an effective treatment for anxiety disorders, including Generalized Anxiety Disorder. It is also well-tolerated by patients. The only side effects that have been identified so far are mild gastrointestinal symptoms (including burping and breath odour) and these are uncommon. The results of a small pilot study suggest that Silexan may also be effective and well-tolerated in PTSD.

The STOP trial is a clinical trial that aims to investigate whether adding Silexan to treatment-as-usual improves PTSD symptoms in adults with PTSD. The trial will recruit 278 participants. Participants will be randomly assigned to take Silexan or a placebo (look-alike dummy pills) daily in addition to their usual medications for 12 weeks. The severity of their PTSD symptoms will be assessed prior to and at the end of this 12-week period.

The STOP trial has the potential to obtain definitive evidence regarding whether Silexan helps treat symptoms of PTSD. If Silexan is found to be an effective treatment for PTSD, the pool of patients who could potentially benefit from this treatment includes any adults with PTSD. Silexan is already available over-the-counter at a relatively low cost so there will be few barriers to accessing this treatment.

DETAILED DESCRIPTION:
Background: Posttraumatic stress disorder (PTSD) is a common and debilitating psychiatric disorder. Existing PTSD treatments have very significant limitations. Current evidence-based treatments for PTSD include trauma-focussed psychotherapy and antidepressant medications, including selective serotonin reuptake inhibitors and the serotonin noradrenaline reuptake inhibitor venlafaxine. Many patients are unable to tolerate trauma-focussed psychotherapy. Uptake is relatively low and dropout rates are high. In addition, up to 50% of patients fail to respond to this therapy. Antidepressant medications have small clinical effects and are associated with unpleasant side effects that can lead to non-adherence. There is an urgent need for new treatments for PTSD that are effective and well-tolerated. Silexan has the potential to provide a transformative alternative to these treatments. It is an orally administered lavender oil preparation whose main constituents are the monoterpenoids linalool and linalyl acetate. It is available over-the-counter in 14 countries, including Australia and the United States. It has a novel pharmacodynamic profile that includes potent inhibition of voltage-gated calcium channels and reduction of serotonin 1A receptor binding potential. Silexan is an effective treatment for Generalized Anxiety Disorder (GAD) and other anxiety disorders. A 2019 independent meta-analysis of data from five randomized controlled trials involving 1,320 participants with anxiety disorders found that Silexan 160 mg out-performed paroxetine and lorazepam in reducing anxiety symptoms. Silexan is also well-tolerated. The only adverse effects that have been identified so far are mild gastrointestinal symptoms and these are uncommon. Promising pilot data suggest that Silexan may also be effective and well-tolerated in PTSD.

Hypothesis: The primary hypothesis is that Silexan, as an adjunct to treatment-as-usual, over 12 weeks will be superior to placebo in improving PTSD symptoms in adults with PTSD.

Specific aims: The trial aims to investigate the effectiveness of adjunctive Silexan, compared with placebo, over 12 weeks in improving PTSD symptoms. The primary outcome measure will be the between-group change from baseline in the total symptom severity score on the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).

Study design: The trial is a phase 3, 12-week, multi-site, parallel-arm, randomized, placebo-controlled, double-blind trial. Participants will be adults with PTSD without comorbid psychosis, bipolar disorder, moderate or severe substance use disorder or Borderline Personality Disorder. Participants randomized to the Silexan arm will receive Silexan 160 mg daily for 12 weeks in addition to their usual prescribed medications. Participants randomized to the placebo arm will receive capsules containing an inert placebo. The target sample size will be 250 participants, or 125 per arm. The study will recruit 278 participants to account for a 10% drop-out rate.

Clinical impact: There is an urgent need to develop new treatments for PTSD that are effective and well-tolerated. This trial has the potential to provide definitive evidence of the efficacy of Silexan in adult PTSD. Silexan is safe, well-tolerated, currently available and affordable, facilitating a rapid translation into clinical care. If Silexan is found to be an effective treatment for PTSD, the pool of patients who could potentially benefit from this treatment includes any adults with PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over.
2. Fluent in English.
3. Meet DSM-5 criteria for PTSD, irrespective of occupation (e.g. first responder, police officer, ex-military or civilian), determined using the Mini International Neuropsychiatric Interview 7.0.2.
4. Have a score on the PTSD Checklist for DSM-5 (PCL-5) equal to or over 33.

Exclusion Criteria:

1. Are currently serving in the Australian Defence Force
2. Lifetime history of a psychotic or bipolar disorder, or dissociative identity disorder.
3. Moderate or severe alcohol or other substance use disorder within 3 months of screening.
4. Active suicidal or homicidal ideation.
5. Borderline Personality Disorder (BPD).
6. Acute or unstable medical illness or other significant medical condition, that would make participation in the trial unsafe or inappropriate.
7. Pregnancy, lactation or unwillingness to use an acceptable method of contraception (required for both males and females who are of reproductive potential and sexually active with partners of the opposite sex) through the duration of participants' involvement in the study up to and including week 16. Participants will also be advised not to donate eggs or sperm during the study period.
8. Commencement of a trauma-focussed psychotherapy (including Prolonged Exposure, Cognitive Processing Therapy and Eye Movement Desensitisation and Reprocessing) within 3 months of screening.
9. Commencement or change in dose of psychoactive medications within 4 weeks of screening.
10. Participants will be asked not to initiate psychotherapy or change the dose of psychoactive medications during the course of the study except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the participant or terminating their participation.
11. Severe acquired brain injury.
12. Individual is not eligible for public mental health services due to their visa status in Australia or for any other reason.
13. Any other condition that in the opinion of the research team is likely to make completion of the trial requirements infeasible.
14. Inability to understand or speak English to the extent necessary to give informed consent and complete the trial (researcher or clinician-determined).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | At baseline and at week 12 of the study period
  The Primary Outcome Measure will be the between-group difference in the change from baseline to week 12 in the total symptom severity score on the CAPS-5. The CAPS-5 has good internal consistency, inter-rater reliability, test-retest reliability and convergent validity in measuring PTSD symptom severity, and is regarded as the gold-standard for measuring PTSD symptoms in research settings. The CAPS-5 will be used to query the presence of PTSD symptoms across the two weeks prior to each CAPS-5 assessment. We will also compare between-group differences in remission rates of PTSD, as determined by the CAPS-5.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of anxiety symptoms on the HAM-A. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Hamilton Anxiety Rating Scale consists of 14 items and is the most widely used interview instrument for measurement of anxiety in adults and children.
Generalized Anxiety Disorder-7 (GAD-7) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of anxiety symptoms on the GAD-7. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Generalized Anxiety Disorder-7 is a 7-item scale with each item scores on a scale of 0 ("not at all") to 3 ("nearly every day") based on symptom presentation in the past two weeks.
Generalized Anxiety Disorder-7 (GAD-7) | At baseline, week 4, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of anxiety symptoms on the GAD-7, measured at baseline, week 4, week 8 and week 12 of treatment. The Generalized Anxiety Disorder-7 is a 7-item scale with each item scores on a scale of 0 ("not at all") to 3 ("nearly every day") based on symptom presentation in the past two weeks.
Beck Depression Inventory-II (BDI-II) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of depressive symptoms on the BDI-II. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The BDI-II comprises of 21 questions rated on 4-point scales of severity (0-3), with a total score that reflects the level or degree of depression. The BDI-II has high internal consistency.
Patient Health Questionnaire-9 (PHQ-9) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of depressive symptoms on the PHQ-9. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Patient Health Questionnaire-9 is a screening measure of depressive symptoms. The PHQ-9 asks participants to rate each of the 9 DSM-IV criteria for major depressive disorder from 0 ("not at all") to 3 ("nearly every day").
Patient Health Questionnaire-9 (PHQ-9) | At baseline, week 4, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of depressive symptoms on the PHQ-9, measured at baseline, week 4, week 8 and week 12 of treatment. The Patient Health Questionnaire-9 is a screening measure of depressive symptoms. The PHQ-9 asks participants to rate each of the 9 DSM-IV criteria for major depressive disorder from 0 ("not at all") to 3 ("nearly every day").
Patient Health Questionnaire-15 (PHQ-15) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of somatic symptoms on the PHQ-15. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Patient Health Questionnaire-15 is a Patient Health Questionnaire module designed to assess the presence of somatic symptoms. The PHQ-15 has good internal consistency and test-retest reliability.
Patient Health Questionnaire-15 (PHQ-15) | At baseline, week 4, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of somatic symptoms on the PHQ-15, measured at baseline, week 4, week 8 and week 12 of treatment. The Patient Health Questionnaire-15 is a Patient Health Questionnaire module designed to assess the presence of somatic symptoms. The PHQ-15 has good internal consistency and test-retest reliability.
Pittsburgh Sleep Quality Index, with Addendum for PTSD (PSQI & PSQI-A) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of sleep quality on the PSQI & PSQI-A. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Pittsburgh Sleep Quality Index is designed to measure overall sleep quality during the previous month in a clinical population. The PSQI comprises 19 questions across 7 domains or "component" scores, each weighted equally on a 0-3 scale. The PSQI will include the PTSD Addendum (PSQI-A), which are 10 additional questions designed to assess the frequency of disruptive nocturnal behaviours.
Pittsburgh Sleep Quality Index, with Addendum for PTSD (PSQI & PSQI-A) | At baseline, week 4, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of sleep quality on the PSQI & PSQI-A, measured at baseline, week 4, week 8 and week 12 of treatment. The Pittsburgh Sleep Quality Index is designed to measure overall sleep quality during the previous month in a clinical population. The PSQI comprises 19 questions across 7 domains or "component" scores, each weighted equally on a 0-3 scale. The PSQI will include the PTSD Addendum (PSQI-A), which are 10 additional questions designed to assess the frequency of disruptive nocturnal behaviours.
Alcohol Use Disorders Identification Test (AUDIT) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of problematic alcohol use on the AUDIT. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Alcohol Use Disorders Identification Test is a 10-item questionnaire developed through a 6-country World Health Organization collaborative project, as a screening tool for harmful alcohol consumption. The AUDIT spans the domains of alcohol consumption, drinking behaviour, and alcohol-related problems that may have occurred in the past year, as well as lifetime exposure.
Alcohol Use Disorders Identification Test (AUDIT) | At baseline, week 4, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of problematic alcohol use on the AUDIT, measured at baseline, week 4, week 8 and week 12 of treatment. The Alcohol Use Disorders Identification Test is a 10-item questionnaire developed through a 6-country World Health Organization collaborative project, as a screening tool for harmful alcohol consumption. The AUDIT spans the domains of alcohol consumption, drinking behaviour, and alcohol-related problems that may have occurred in the past year, as well as lifetime exposure.
World Health Organization (WHO) Disability Assessment Schedule (WHODAS 2.0) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of functional disability on the WHODAS 2.0. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The 12-item self-report version of the World Health Organization (WHO) Disability Assessment Schedule is a measure of functioning and disability across six major life domains due to health conditions. The WHODAS has high internal consistency and test-retest reliability.
General Well Being Schedule (GWBS) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of general well-being on the GWBS. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The General Well Being Schedule is an 18-item measure of subjective psychological well-being and distress. The GWBS has good test-retest reliability, as well as internal consistency for both sexes.
Assessment of Quality of Life-6D (AQoL-6D) | At baseline, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the between-group difference in the change from baseline to week 12, and baseline to week 16 (while including all available time-points including the off-treatment period) in measures of quality of life on the AQoL-6D. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The Assessment of Quality of Life-6D scale is a 20-item, 6-dimensional measure with each item containing between 4 and 6 response levels. The AQoL-6D assesses the following 6 domains of quality of life: Independent Living, Relationships, Mental Health, Coping, Pain and Senses.
PTSD Checklist for DSM-5 (PCL-5) | At intake, at week 12 and at week 16 of the study period
  One of the Secondary Outcome Measures will be the will be the between-group difference in the change from intake to week 12, and intake to week 16 (while including all available time-points including the off-treatment period) in measures of quality of life on the PCL-5. Additional comparisons for between-group differences from week 12 to week 16 will also be performed. The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and intensity of each of the 20 DSM-5 PTSD symptoms. The PCL-5 has been shown to have strong reliability and validity. A score of ≥ 33 suggests PTSD.
PTSD Checklist for DSM-5 (PCL-5) | At intake, week 2, week 4, week 6, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of PTSD symptom severity on the PCL-5, measured at intake, and at week 2, week 4, week 6, week 8 and week 12 of treatment. The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and intensity of each of the 20 DSM-5 PTSD symptoms. The PCL-5 has been shown to have strong reliability and validity. A score of ≥ 33 suggests PTSD.
Patient Global Impression of Change Scale (PGIC) | Week 2, week 4, week 6, week 8 and week 12 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of patient global impression of change on the PGIC, measured at week 2, week 4, week 6, week 8 and week 12 of treatment. The Patient Global Impression of Change Scale asks participants to rate the change (if any) that they have experienced since starting treatment, on a scale of 1 ("No change") to 7 ("A great deal better and a considerable improvement that has made all the difference").
Actigraphy watches | Continously from baseline until week 16 of the study period
  One of the Secondary Outcome Measures will be the longitudinal trajectory analysis of sleep, actigraphy, and physiological measures (including mean heart rate, mean heart rate variability, mean blood pressure), measured continuously throughout the study period (baseline to week 16).

OTHER OUTCOMES:
Mediators of response to Silexan | Baseline
  We will assess whether additional pre-existing factors, including social support (measured via the Social Support Survey (SSS)), past military deployment (measured via the Deployment Risk & Resilience Inventory-2 (DRRI-2)), or developmental trauma (measured via the BRFSS Adverse Childhood Experience (ACE) Module) affect response to Silexan.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berk, PhD, Principal Investigator — Deakin University
Locations (4):
- Australia (4):
  - University of Melbourne, Carlton, Victoria
  - Deakin University, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Ramsay Clinic Albert Road, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The National Institute of Mental Health Data Archive (NDA) will be used as an online data-sharing repository. De-identified participant data will be linked in the shared data repository using an assigned NDA Global Unique Identifier (GUID). The GUID itself is not personally identifiable information or protected health information.
Supporting Information: ICF
Time Frame: A copy of the blank, ethics-approved consent form will be posted on clinicaltrials.gov, after the trial is closed to recruitment and no later than 60 days after the last study visit, in accordance with United States federal requirements described in Code of Federal Regulations, Title 32, Part 219 (32 CFR 219).
URL: https://nda.nih.gov/